CLINICAL TRIAL: NCT02276924
Title: Diagnostic Relevance of Laser Confocal Microscopy During Reno-ureteroscopy in the Context of the Screening and Follow-up of Upper Urinary Tract Tumors
Brief Title: Diagnostic Relevance of Laser Confocal Microscopy for the Screening of Upper Urinary Tract Tumors
Acronym: UROVISIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0026
Record Dates: First submitted 2014-08-29; First posted 2014-10-28 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hematuria; Nephrolithiasis; Cancer of Urinary Tract; Ureteropelvic Junction Obstruction
Keywords: Laser Confocal Microscopy; Superior Urinary Tract Tumors
MeSH Terms: conditions — Hematuria; Nephrolithiasis; Urologic Neoplasms; Multicystic renal dysplasia, bilateral | interventions — Microscopy, Confocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser confocal microscopy (Experimental): Patients undergoing a reno-ureteroscopy for diagnosis or treatment indication will follow a laser confocal microscopy procedure.
  Interventions: Device: Laser confocal microscopy

INTERVENTIONS:
Device: Laser confocal microscopy — Patients undergoing a reno-ureteroscopy for diagnosis or treatment indication will receive an intra-vesical instillation of fluorescein (0.1%) for 5 minutes, followed by the laser confocal microscopy procedure.
  Other Names: Cell-vizio

SUMMARY:
Upper Urinary Tract Tumors have an incidence of 1 to 2 cases for 100 000 persons per year. The standard treatment for these tumors is the ablation of the kidney, ureter and a part of the bladder surrounding the ureteral orifice. The development of new diagnosis and treatment techniques through natural routes opens the possibility to use conservative treatments. The investigators hypothesis is that during a reno-ureteroscopy, laser confocal microscopy will allow the discrimination between normal and pathologic urothelium by microscopic analysis. This will prevent the systematic use of biopsies which are often difficult and iatrogenic.

DETAILED DESCRIPTION:
The objective of the present study is to assess contribution of laser confocal microscopy in diagnosing of upper urinary tract tumors during a reno-uteroscopy compared to analysing of architectural elements (vascular characteristics, organization) and cellular (morphology, cohesion, border).

ELIGIBILITY:
Inclusion Criteria:

* Any legally adult fully informed patient who consent to participate to the study
* Patient followed by the Urology Department
* Indication for a diagnosis or treatment reno-ureteroscopy
* Coverage of the social insurance

Exclusion Criteria:

* Minor Patient
* Pregnancy or breast feeding
* Concomitant treatment (for example beta-blocker)
* Contra-indication to general anaesthesia
* Hypersensitivity to sodium fluorescein
* Medical history of cardio-pulmonary disease (myocardial infarction, cardiovascular event, bronchospasm ...) due to fluorescein instillation
* Medical history of asthma or allergy due to fluorescein instillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic relevance of laser confocal microscopy compared to the cytological and histological data, during reno-ureteroscopy according to Chang's reference criteria | 24 months
  According to Chang's reference criteria, we will define the urothelial microarchitecture (normal, papillary, inflammatory, low grade lesion, high grade lesion, in situ carcinoma). The diagnostic relevance of the MCL (absence or presence of the lesion) will be compare to the reference tests calculating sensibility, specificity and predictive values

SECONDARY OUTCOMES:
Inter- and intra-observer diagnostic concordance | 24 months
  Anonymized videos of the intervention will be reviewed at the end of the study by a "naive" surgeon to assess inter-observer concordance. A concordance Kappa test will be performed
Surgery duration | 24 months
Reference atlas | 24 months
  Videos and images quality will be assessed to compile them in a refence atlas

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Bonnal, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille, Hauts-de-France, France

REFERENCES:
- [Result] Marien A, Rock A, Maadarani KE, Francois C, Gosset P, Mauroy B, Bonnal JL. Urothelial Tumors and Dual-Band Imaging: A New Concept in Confocal Laser Endomicroscopy. J Endourol. 2017 May;31(5):538-544. doi: 10.1089/end.2016.0892. Epub 2017 Mar 22. PMID 28326794